CLINICAL TRIAL: NCT03529747
Title: Exploring the Effectiveness of Online Self-help for Parents of Children With Food Allergies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canterbury Christ Church University (Other)
Collaborators: Brighton & Sussex Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NaomiSugunasinghaMRP2017
Record Dates: First submitted 2018-05-08; First posted 2018-05-18 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2019-10

CONDITIONS: The Well Being of Parents of Children With Food Allergies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online self-help (Experimental): A website providing information and psycho-education aimed at parents and carers of children with food allergies.
  Interventions: Other: Online self-help
- Wait list control (No Intervention): A waiting list control group, who will receive access to the online self-help once the RCT is complete.

INTERVENTIONS:
Other: Online self-help — As detailed in experimental arm description.
  Arms: Online self-help

SUMMARY:
This study aims to conduct an initial evaluation of whether online self-help can improve the quality of life of parents of children with food allergies.

DETAILED DESCRIPTION:
This study is a pilot randomised controlled trial (RCT) comparing online self-help for parents of children with food allergies with a wait-list control. A battery of self-report measures will be administered online at baseline (week 0), post-intervention (week 4) and at follow-up (week 8).

ELIGIBILITY:
Inclusion Criteria:

* Being a parent of at least one child (under the age of 18) who has a food allergy.
* Adequate understanding of written English.

Exclusion Criteria:

* Having consulted on the design of the self-help website.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2019-02-04 (Actual); Study Completion 2019-02-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline at 4-weeks on the Food Allergy Quality of Life Parental Burden scale | Post-intervention (4-weeks after baseline)
  This measures parental burden when caring for a food-allergic child, producing a score between 17 and 119, with higher scores indicating greater burden.

SECONDARY OUTCOMES:
Change from baseline at 8-weeks on the Food Allergy Quality of Life Parental Burden scale | Follow-up (8-weeks after baseline)
  This measures parental burden when caring for a food-allergic child, producing a score between 17 and 119, with higher scores indicating greater burden.
Change from baseline at 4-weeks on the Patient Health Questionnaire depression scale 8 | Post-intervention (4-weeks after baseline)
  This measures symptoms of depression, producing a score between 0 and 24, with higher scores indicating greater symptomatology.
Change from baseline at 8-weeks on the Patient Health Questionnaire depression scale 8 | Follow-up (8-weeks after baseline)
  This measures symptoms of depression, producing a score between 0 and 24, with higher scores indicating greater symptomatology.
Change from baseline at 4-weeks on the Generalised Anxiety Disorder 7 scale | Post-intervention (4-weeks after baseline)
  This measures symptoms of generalised anxiety disorder, producing a score between 0 and 21, with higher scores indicating greater symptomatology.
Change from baseline at 8-weeks on the Generalised Anxiety Disorder 7 scale | Follow-up (8-weeks after baseline)
  This measures symptoms of generalised anxiety disorder, producing a score between 0 and 21, with higher scores indicating greater symptomatology.
Change from baseline at 4-weeks on the Perceived Stress Scale (10 items) | Post-intervention (4-weeks after baseline)
  This produces a score between 0 and 40, with higher scores indicating higher levels of perceived stress.
Change from baseline at 8-weeks on the Perceived Stress Scale (10 items) | Follow-up (8-weeks after baseline)
  This produces a score between 0 and 40, with higher scores indicating higher levels of perceived stress.

OTHER OUTCOMES:
Change from baseline at 4-weeks on the Food Allergy Self-Efficacy Scale for Parents | Post-intervention (4-weeks after baseline)
  This measures a parent's confidence in managing their child's food allergy, producing a score between 0 and 100, with higher scores indicating greater confidence.
Change from baseline at 8-weeks on the Food Allergy Self-Efficacy Scale for Parents | Follow-up (8-weeks after baseline)
  This measures a parent's confidence in managing their child's food allergy, producing a score between 0 and 100, with higher scores indicating greater confidence.
Change from baseline at 4-weeks on the Intolerance of Uncertainty Scale | Post-intervention (4-weeks after baseline)
  This measures participants' ability to tolerate uncertainty, producing scores between 27 and 135, with higher scores indicating lower tolerance of uncertainty.
Change from baseline at 8-weeks on the Intolerance of Uncertainty Scale | Follow-up (8-weeks after baseline)
  This measures participants' ability to tolerate uncertainty, producing scores between 27 and 135, with higher scores indicating lower tolerance of uncertainty.

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Sugunasingha, BSc, PGCert, Principal Investigator — Canterbury Christ Church University; Fergal Jones, PhD, PsychD, Study Director — Canterbury Christ Church University; Christina Jones, PhD, Study Director — Brighton & Sussex Medical School
Locations (1):
- Salomons Centre for Applied Psychology, Canterbury Christ Church University, Royal Tunbridge Wells, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided